CLINICAL TRIAL: NCT01952665
Title: A Multi-Center Study Comparing the Clinical Performance of Two Silicone Hydrogel Lenses Over 1 Month of Daily Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EX-MKTG-41
Record Dates: First submitted 2013-09-18; First posted 2013-09-30 (Estimated); Results first posted 2015-09-24 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-05

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- comfilcon A (Active Comparator): Daily wear soft contact lens comfilcon A
  Interventions: Device: lotrafilcon B
- lotrafilcon B (Active Comparator): Daily wear soft contact lens lotrafilcon B
  Interventions: Device: comfilcon A

INTERVENTIONS:
Device: comfilcon A — Each subject randomized to wear the test lens (comfilcon A) or the control lens (lotrafilcon B) for one month of daily wear before repeating schedule for the second pair without a washout period.
  Arms: lotrafilcon B
Device: lotrafilcon B — Each subject randomized to wear the test lens (comfilcon A) or the control lens (lotrafilcon B) for one month of daily wear before repeating schedule for the second pair without a washout period.
  Arms: comfilcon A

SUMMARY:
A Multi-Center Study Comparing the Clinical Performance of Two Silicone Hydrogel Lenses Over 1 Month of Daily Wear

DETAILED DESCRIPTION:
Two-month, single masked, randomized, bilateral, crossover, 1-month of daily wear in each study lens.

ELIGIBILITY:
Inclusion Criteria:

* Is between 18 and 40 years of age (inclusive)
* Have the use of a mobile phone to send and receive text messages throughout the day for the duration of the study
* Has had a self-reported visual exam in the last two years
* Is an adapted soft CL wearer
* Has a Contact Lens (CL) spherical prescription between - 1.00 and - 9.00 (inclusive)
* Has less than 0.75D spectacle cylinder in each eye
* Is correctable to a visual acuity of 20/25 or better in both eyes
* Has clear corneas and no active ocular disease
* Has read, understood and signed the information consent letter
* Is willing to comply with the wear schedule (at least 40 hrs per week)
* Is willing to comply with the visit schedule

Exclusion Criteria:

* Has never worn contact lenses before
* Currently wears rigid gas permeable contact lenses
* Has a history of not achieving comfortable CL wear (5 days per week; > 8 hours/day)
* Has a contact lens prescription outside the range of - 1.00 to -9.00D
* Has a spectacle cylinder greater than -0.50D of cylinder in either eye
* Has best corrected spectacle distance vision worse then 20/25 in either eye
* Has any systemic disease affecting ocular health
* Is using any systemic or topical medications that will affect ocular health
* Has any ocular pathology or severe insufficiency of lacrimal secretion
* Has persistent, clinically significant corneal or conjunctival staining
* Has active neovascularization or any central corneal scars
* Is aphakic
* Is presbyopic
* Has undergone corneal refractive surgery
* Is participating in any other type of eye related clinical or research study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Siegel, OD, Principal Investigator — CooperVision, US
Locations (6):
- United States (6):
  - Family Eye Care Center, Campbell, California
  - Golden Optometric Group, Whittier, California
  - Drs. Quinn, Foster, &Associates, Athens, Georgia
  - Davis EyeCare Associates, Oak Lawn, Illinois
  - Kannarr Eye Care LLC, Pittsburg, Kansas
  - Complete Eye Care of Medina, Medina, Minnesota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 1 month, cross-over dispensing study conducted at 6 clinical sites in the US. 63 subjects were enrolled, 12 were discontinued and 51 completed the study.
Groups:
- Comfilcon A Then Lotrafilcon B; Lotrafilcon B Then Comfilcon A: Each subject randomized to wear either the test lens (comfilcon A) or the control lens (lotrafilcon B) for one month of daily wear before repeating schedule for the second pair without a washout period.
Period: Overall Study
Arm/Group | Comfilcon A Then Lotrafilcon B | Lotrafilcon B Then Comfilcon A
Started | 37 | 26
Completed | 31 | 20
Not Completed | 6 | 6
Not completed — Physician Decision | 3 | 2
Not completed — Lost to Follow-up | 1 | 2
Not completed — Adverse Event | 2 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Comfilcon A Then Lotrafilcon B; Lotrafilcon B Then Comfilcon A: Each subject randomized to wear the test lens (comfilcon A) or the control lens (lotrafilcon B) for one month of daily wear before repeating schedule for the second pair without a washout period.
- Total: Total of all reporting groups
Arm/Group | Comfilcon A Then Lotrafilcon B | Lotrafilcon B Then Comfilcon A | Total
Number analyzed (Participants) | 37 | 26 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 26 | 63
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 15 | 38
  Male | 14 | 11 | 25
Region of Enrollment [Number; unit: participants]
  United States | 37 | 26 | 63

OUTCOME MEASURES:

1. Primary Outcome: Comfort at Insertion
Description: Participant rating for lens comfort on insertion. Collected at dispense for both study lens pairs. (0-10, 0= Very Uncomfortable, 10= Cannot feel).
Time Frame: Dispense
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 63 | 60
units on a scale | 9.21 (1.06) | 8.22 (1.98)

2. Primary Outcome: Visual Quality
Description: Participant rating of visual quality. Collected at dispense for both study pairs. (0-10, 0= Very Poor Vision, 10= Perfectly Sharp, Clear Vision)
Time Frame: Dispense
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 63 | 60
units on a scale | 9.27 (1.02) | 8.87 (1.89)

3. Secondary Outcome: Binocular Visual Acuity logMAR
Description: Assessment of visual acuity (VA). Collected at 2 weeks for both study lens pairs. Binocular High Contrast Distance. logMAR (negative logMAR values indicates better Visual Acuity (VA)). 0.0 logMAR = 20/20 snellen chart
Time Frame: Dispense
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 63 | 60
logMAR | -0.052 (0.048) | -0.054 (0.050)

4. Secondary Outcome: Surface Wetting
Description: Assessment of surface wetting by slit lamp. Collected at dispense for both study pairs. 0=Non-wettable surface, 1= > 1 non-wetting area of some magnitude., 2=One non-wetting area of some magnitude, 3=Hazy surface that resolves with a blink. Typical soft lens appearance with long drying time., 4=Smooth uniformly reflective surface. Appearance of a healthy cornea (Grade 0-4 in ½ steps)
Time Frame: Dispense
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 63 | 60
Number analyzed (eyes) | 126 | 120
units on a scale | 7.59 (1.45) | 7.75 (1.09)

5. Secondary Outcome: Surface Deposition
Description: Assessment of surface deposition by slit lamp. Collected at dispense for both study pairs. (Grade 0-4 in ½ steps; Clean= 0; Deposited = 4)
Time Frame: Dispense
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 63 | 60
Number analyzed (eyes) | 126 | 120
units on a scale | 0.37 (1.46) | 0.23 (1.10)

6. Secondary Outcome: Centration
Description: Assessment of lens centration. Collected at dispense for both study pairs. Biomicroscopy; by degree and direction in the primary position. (Rated as Optimal Centration or Not Optimal)
Time Frame: Dispense
Measure: Number; unit: lenses
Units Other Than Participants: lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 63 | 60
Number analyzed (lenses) | 126 | 120
lenses
  Optimal Centration | 116 | 109
  Not Optimal Centration | 10 | 11

7. Secondary Outcome: Corneal Coverage
Description: Assessment of lens corneal coverage. Collected at dispense for both study pairs. Biomicroscopy; assessed in primary gaze. (Rated as Normal Coverage or Not Covering)
Time Frame: Dispense
Measure: Number; unit: lenses
Units Other Than Participants: lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 63 | 60
Number analyzed (lenses) | 126 | 120
lenses
  Normal Coverage | 126 | 118
  Not Covering | 0 | 2

8. Secondary Outcome: Post Blink Movement
Description: Assessment of post blink movement. Collected at dispense for both study lens pairs. Assessed immediately after the blink. (0-4, 0=Insufficient, unacceptable movement, 1=Minimal, but acceptable movement, 2=Optimal movement, 3=Moderate, but acceptable movement, 4=Excessive, unacceptable movement)
Time Frame: Dispense
Measure: Number; unit: lenses
Units Other Than Participants: lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 63 | 60
Number analyzed (lenses) | 126 | 120
lenses
  Movement Grade 0 | 0 | 0
  Movement Grade 1 | 11 | 13
  Movement Grade 2 | 104 | 92
  Movement Grade 3 | 11 | 15
  Movement Grade 4 | 0 | 0

9. Secondary Outcome: Push Up Test
Description: Assessment of lens tightness. Collected at dispense for both study pairs. Digital push up test. Continuous Scale (0-100%, 0%=Falls from cornea without lid support, 50%= Optimum, 100%= No movement)
Time Frame: Dispense
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 60 | 63
Number analyzed (lenses) | 120 | 126
units on a scale | 49.25 (11.42) | 48.13 (11.34)

10. Secondary Outcome: Overall Fit Acceptance
Description: Assessment of overall lens fit acceptance. Collected at dispense for both study pairs. (0-4, 0=should not be worn, 1=borderline but unacceptable, 2=minimally acceptable, early review, 3=not perfect but okay to dispense, 4=perfect)
Time Frame: Dispense
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 63 | 60
Number analyzed (lenses) | 126 | 120
units on a scale | 3.74 (0.48) | 3.68 (0.47)

11. Other Pre Specified Outcome: The Number of Trials Needed to Achieve Final Dispensing Pair of Study Lenses.
Description: The number of trials needed to achieve final dispensing pair of study lenses. Number of lenses required to dispense the final pair of study lenses. Collected at dispense for both study lens pairs. (Number required; 1, 2, 3, >3)
Time Frame: Dispense
Measure: Mean (Standard Deviation); unit: number of trial lenses
Units Other Than Participants: lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 63 | 60
Number analyzed (lenses) | 126 | 120
number of trial lenses | 2.06 (0.30) | 2.03 (0.18)

12. Primary Outcome: Average Daily Wearing Time
Description: Participants measure of average daily wear time for study lenses at 2 Weeks.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 58 | 57
hours | 13.72 (2.66) | 13.82 (2.95)

13. Secondary Outcome: Rewetting Drops
Description: Participant use of rewetting drops. Collected at 2 weeks for both study lens pairs. (Uses rewetting drops / Does not use rewetting drops).
Time Frame: 2 weeks
Measure: Number; unit: participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 58 | 57
participants
  Uses | 50 | 47
  Does Not Use | 8 | 10

14. Primary Outcome: Comfortable Wearing Time
Description: Participant rating of lens Comfortable Wearing Time for both study pairs. After 2 weeks wear for each pair. (The hours of average comfortable wearing time)
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 58 | 57
hours | 11.07 (3.87) | 11.14 (3.72)

15. Primary Outcome: Comfort
Description: Participant rating for lens comfort. After 2 weeks wear for each study pair. (0-10, 0= Very Uncomfortable, 10= Cannot Feel).
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 58 | 57
units on a scale
  Insertion | 8.78 (1.48) | 8.35 (1.68)
  During Day | 8.29 (1.63) | 8.09 (1.76)
  Prior to Removal | 7.31 (2.20) | 7.00 (1.95)
  Overall | 8.28 (1.58) | 7.84 (1.75)

16. Primary Outcome: Dryness
Description: Participant rating for lens dryness. After 2 weeks wear for each study pair. (0-10, 0= Very Dry, 10= No Dryness).
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 58 | 57
units on a scale
  During Day | 8.19 (1.76) | 7.95 (1.71)
  Prior to Removal | 7.21 (2.27) | 6.89 (1.93)
  Overall | 7.97 (1.90) | 7.60 (1.70)

17. Primary Outcome: Handling
Description: Participant rating for lens handling. After 2 weeks wear for each study pair. (0-10, 0= Very Difficult, 10= Very Easy).
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 58 | 57
units on a scale
  Insertion/Removal | 9.19 (1.48) | 9.37 (0.90)
  Overall | 9.21 (1.42) | 9.39 (0.90)

18. Primary Outcome: Vision Satisfaction
Description: Participant rating for vision satisfaction. After 2 weeks wear for each study pair. (0-10, 0= Very Unsatisfied, 10= Very Satisfied)
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 58 | 57
units on a scale | 9.10 (1.83) | 8.82 (1.69)

19. Primary Outcome: Eye Whiteness/Redness
Description: Participant rating for Eye Whiteness/Redness. After 2 weeks wear for each study pair. (0-10, 0= Significant Redness, 10= Totally White)
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 58 | 57
units on a scale | 8.69 (1.90) | 8.72 (1.61)

20. Primary Outcome: Overall Sensation of Moistness
Description: Participant rating of overall sensation for moistness (hydration). After 2 weeks wear for each study pair. 5-point Likert Scale; 1=Excellent, 2=Good, 3=Average, 4=Below Average, 5=Poor.
Time Frame: 2 weeks
Measure: Number; unit: participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 58 | 57
participants
  Excellent | 17 | 12
  Good | 25 | 24
  Average | 9 | 12
  Fair | 6 | 7
  Poor | 1 | 2

21. Primary Outcome: Overall Sensation of Smoothness
Description: Participant rating of overall sensation for smoothness (deposit resistance). After 2 weeks wear for each study pair. 5-point Likert Scale; 1=Excellent, 2=Good, 3=Average, 4=Below Average, 5=Poor.
Time Frame: 2 weeks
Measure: Number; unit: participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 58 | 57
participants
  Excellent | 23 | 21
  Good | 17 | 20
  Average | 13 | 12
  Fair | 5 | 1
  Poor | 0 | 3

22. Primary Outcome: Overall Comfort Satisfaction
Description: Participant rating of satisfaction regarding comfort. After 2 weeks wear for each study pair. 4-point Likert Scale; 1=Completely Satisfied, 2=Somewhat Satisfied, 3=Somewhat Dissatisfied, 4=Completely Dissatisfied
Time Frame: 2 weeks
Measure: Number; unit: participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 58 | 57
participants
  Completely Satisfied | 30 | 20
  Somewhat Satisfied | 18 | 26
  Somewhat Dissatisfied | 9 | 7
  Completely Dissatisfied | 1 | 4

23. Primary Outcome: Overall Dryness Satisfaction
Description: Participant rating of satisfaction regarding dryness. After 2 weeks wear for each study pair. 4-point Likert Scale; 1=Completely Satisfied, 2=Somewhat Satisfied, 3=Somewhat Dissatisfied, 4=Completely Dissatisfied
Time Frame: 2 weeks
Measure: Number; unit: participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 58 | 57
participants
  Completely Satisfied | 24 | 20
  Somewhat Satisfied | 23 | 22
  Somewhat Dissatisfied | 9 | 11
  Completely Dissatisfied | 2 | 4

24. Primary Outcome: Overall Handling Satisfaction
Description: Participant rating of satisfaction regarding handling. After 2 weeks wear for each study pair. 4-point Likert Scale; 1=Completely Satisfied, 2=Somewhat Satisfied, 3=Somewhat Dissatisfied, 4=Completely Dissatisfied
Time Frame: 2 weeks
Measure: Number; unit: participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 58 | 57
participants
  Completely Satisfied | 49 | 43
  Somewhat Satisfied | 6 | 13
  Somewhat Dissatisfied | 3 | 1
  Completely Dissatisfied | 0 | 0

25. Primary Outcome: Overall Vision Satisfaction
Description: Participant rating of satisfaction regarding vision. After 2 weeks wear for each study pair. 4-point Likert Scale; 1=Completely Satisfied, 2=Somewhat Satisfied, 3=Somewhat Dissatisfied, 4=Completely Dissatisfied
Time Frame: 2 weeks
Measure: Number; unit: participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 58 | 57
participants
  Completely Satisfied | 43 | 35
  Somewhat Satisfied | 12 | 14
  Somewhat Dissatisfied | 1 | 5
  Completely Dissatisfied | 2 | 3

26. Primary Outcome: Overall Satisfaction
Description: Participant rating of satisfaction overall. After 2 weeks wear for each study pair. 4-point Likert Scale; 1=Completely Satisfied, 2=Somewhat Satisfied, 3=Somewhat Dissatisfied, 4=Completely Dissatisfied
Time Frame: 2 weeks
Measure: Number; unit: participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 58 | 57
participants
  Completely Satisfied | 30 | 20
  Somewhat Satisfied | 18 | 26
  Somewhat Dissatisfied | 9 | 7
  Completely Dissatisfied | 1 | 4

27. Primary Outcome: Lens Preference, Pair 1 Comfilcon A
Description: Participant preference for habitual lenses or study lenses with regard to comfort, dryness, handling, vision and overall. Collected at 2 weeks for study pair 1. (Randomized to comfilcon A as pair 1; Forced choice: Pair 1 or Habitual)
Time Frame: 2 weeks
Measure: Number; unit: participants
Groups:
- Habitual Lenses: Subjects attended baseline visit wearing habitual lenses prior to dispense of study lens.
Arm/Group | Comfilcon A | Habitual Lenses
Number analyzed (Participants) | 58 | 58
participants
  Comfort | 26 | 32
  Dryness | 26 | 32
  Handling | 29 | 29
  Vision | 27 | 31
  Overall | 26 | 32

28. Secondary Outcome: Binocular Visual Acuity logMAR
Description: as for outcome 3
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 58 | 57
logMAR | -0.036 (0.076) | -0.037 (0.048)

29. Secondary Outcome: Surface Wetting
Description: Assessment of surface wetting by slit lamp. Collected at 2 weeks for both study lens pairs. 0=Non-wettable surface, 1= > 1 non-wetting area of some magnitude., 2=One non-wetting area of some magnitude, 3=Hazy surface that resolves with a blink. Typical soft lens appearance with long drying time., 4=Smooth uniformly reflective surface. Appearance of a healthy cornea (Grade 0-4 in ½ steps)
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 58 | 57
units on a scale | 7.23 (1.83) | 7.05 (1.61)

30. Secondary Outcome: Surface Deposition
Description: Assessment of surface deposition by slit lamp. Collected at 2 weeks for both study lens pairs. (Grade 0-4 in 1/2 steps; 0=clean, 4=deposited)
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 58 | 57
Number analyzed (eyes) | 116 | 114
units on a scale | 0.46 (0.85) | 1.05 (1.62)

31. Secondary Outcome: Centration
Description: Assessment of lens centration. Collected at 2 weeks. Biomicroscopy; by degree and direction in the primary position. Optimal versus not optimal
Time Frame: 2 Weeks
Measure: Number; unit: lenses
Units Other Than Participants: lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 58 | 57
Number analyzed (lenses) | 116 | 114
lenses
  Optimal Centration | 110 | 100
  Not Optimal Centration | 6 | 14

32. Secondary Outcome: Corneal Coverage
Description: Assessment of lens corneal coverage. Collected at 2 weeks for both study pairs. Biomicroscopy; assessed in primary gaze. (Rated as Normal Coverage or Not Covering)
Time Frame: 2 Weeks
Measure: Number; unit: lenses
Units Other Than Participants: lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 58 | 57
Number analyzed (lenses) | 116 | 114
lenses
  Normal Coverage | 116 | 113
  Not Covering | 0 | 1

33. Secondary Outcome: Post Blink Movement
Description: Assessment of post blink movement. Collected at 2 weeks for both study lens pairs. Assessed immediately after the blink. (Graded 0-4, 0=Insufficient, unacceptable movement, 1=Minimal, but acceptable movement, 2=Optimal movement, 3=Moderate, but acceptable movement, 4=Excessive, unacceptable movement)
Time Frame: 2 Weeks
Measure: Number; unit: lenses
Units Other Than Participants: lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 58 | 57
Number analyzed (lenses) | 116 | 114
lenses
  Movement Grade 0 | 0 | 0
  Movement Grade 1 | 9 | 18
  Movement Grade 2 | 107 | 83
  Movement Grade 3 | 0 | 12
  Movement Grade 4 | 0 | 1

34. Secondary Outcome: Push Up Test
Description: Assessment of lens tightness. Collected at 2 weeks for both study pairs. Digital push up test. (Continuous Scale 0-100%, 0%=Falls from cornea without lid support, 50%= Optimum, 100%= No movement)
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 58 | 57
Number analyzed (lenses) | 116 | 114
units on a scale | 50.78 (10.71) | 51.9 (11.66)

35. Secondary Outcome: Overall Fit Acceptance
Description: Assessment of overall lens fit acceptance. Collected at 2 weeks for both study pairs. (0-4, 0=should not be worn, 1=borderline but unacceptable, 2=minimally acceptable, early review, 3=not perfect but OK to dispense, 4=perfect)
Time Frame: 2 Weeks
Measure: Number; unit: lenses
Units Other Than Participants: lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 58 | 57
Number analyzed (lenses) | 116 | 114
lenses
  Grade 0 | 0 | 0
  Grade 1 | 0 | 2
  Grade 2 | 0 | 0
  Grade 3 | 22 | 41
  Grade 4 | 94 | 71

36. Primary Outcome: Lens Preference, Pair 1 Lotrafilcon B
Description: Participant preference for habitual lenses or study lenses with regard to comfort, dryness, handling, vision and overall. Collected at 2 weeks for study pair 1. (Randomized to lotrafilcon B as pair 1; Forced choice: Pair 1 or Habitual )
Time Frame: 2 weeks
Measure: Number; unit: participants
Arm/Group | Lotrafilcon B | Habitual Lenses
Number analyzed (Participants) | 57 | 57
participants
  Comfort | 19 | 38
  Dryness | 18 | 39
  Handling | 25 | 32
  Vision | 23 | 31
  Overall | 19 | 38

37. Primary Outcome: Comfortable Wearing Time
Description: Participant rating of lens Comfortable Wearing Time for both study pairs. Collected at 4 weeks wear. (The hours of average comfortable wearing time)
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 57 | 56
hours | 11.07 (3.33) | 10.67 (4.15)

38. Primary Outcome: Average Daily Wearing Time
Description: Participants measure of average daily wear time for study lenses at 4 weeks.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 57 | 56
hours | 13.57 (2.88) | 13.91 (2.82)

39. Primary Outcome: Rewetting Drops
Description: Participant use of rewetting drops. Collected at 4 weeks wear for both study lens pairs. (Uses rewetting drops / Does not use rewetting drops).
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 56 | 57
participants
  Uses | 46 | 48
  Does Not Use | 10 | 9

40. Primary Outcome: Comfort
Description: Participant rating for lens comfort. Collected at 4 weeks wear for both study lens pairs. (0-10, 0= Very Uncomfortable, 10= Cannot Feel).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 56 | 57
units on a scale
  Insertion | 8.70 (1.62) | 8.12 (1.83)
  During Day | 8.29 (1.79) | 7.77 (1.80)
  Prior to Removal | 7.38 (2.00) | 6.58 (2.20)
  Overall | 8.07 (1.79) | 7.56 (1.87)

41. Primary Outcome: Dryness
Description: Participant rating for lens dryness. Collected at 4 weeks wear for both study lens pairs. (0-10, 0= Very Dry, 10= No Dryness).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 56 | 57
units on a scale
  During Day | 8.34 (1.72) | 7.70 (2.04)
  Prior to Removal | 7.38 (1.77) | 6.74 (2.31)
  Overall | 8.04 (1.79) | 7.39 (2.05)

42. Primary Outcome: Handling
Description: Participant rating for lens handling. Collected at 4 weeks. (0-10, 0= Very Difficult, 10= Very Easy).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 56 | 57
units on a scale
  Insertion/Removal | 9.21 (1.26) | 9.25 (1.31)
  Overall | 9.27 (1.17) | 9.25 (1.31)

43. Primary Outcome: Vision Satisfaction
Description: Participant rating for vision satisfaction. Collected at 4 weeks wear for both study lens pairs. (0-10, 0= Very Unsatisfied, 10= Very Satisfied)
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 56 | 57
units on a scale | 9.13 (1.60) | 8.51 (1.94)

44. Primary Outcome: Eye Whiteness/Redness
Description: Participant rating for Eye Whiteness/Redness. Collected at 4 weeks wear for both study lens pairs. (0-10, 0= Significant Redness, 10= Totally White)
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 56 | 57
units on a scale | 8.93 (1.28) | 8.53 (1.91)

45. Primary Outcome: Overall Sensation of Moistness
Description: Participant rating of overall sensation for moistness (hydration). Collected at 4 weeks wear for both study lens pairs. 5-point Likert Scale; 1=Excellent, 2=Good, 3=Average, 4=Below Average, 5=Poor.
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 56 | 57
participants
  Excellent | 17 | 13
  Good | 25 | 21
  Average | 9 | 14
  Fair | 4 | 6
  Poor | 1 | 3

46. Primary Outcome: Overall Sensation of Smoothness
Description: Participant rating of overall sensation for smoothness (deposit resistance). Collected at 4 weeks wear for both study lens pairs. 5-point Likert Scale; 1=Excellent, 2=Good, 3=Average, 4=Below Average, 5=Poor.
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 56 | 57
participants
  Excellent | 22 | 18
  Good | 23 | 16
  Average | 8 | 16
  Fair | 3 | 6
  Poor | 0 | 1

47. Primary Outcome: Overall Comfort Satisfaction
Description: Participant rating of satisfaction regarding comfort. Collected at 4 weeks wear for both study lens pairs. 4-point Likert Scale; 1=Completely Satisfied, 2=Somewhat Satisfied, 3=Somewhat Dissatisfied, 4=Completely Dissatisfied
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 56 | 57
participants
  Completely Satisfied | 28 | 20
  Somewhat Satisfied | 21 | 25
  Somewhat Dissatisfied | 5 | 8
  Completely Dissatisfied | 2 | 4

48. Primary Outcome: Overall Dryness Satisfaction
Description: Participant rating of satisfaction regarding dryness. Collected at 4 weeks wear for both study lens pairs. 4-point Likert Scale; 1=Completely Satisfied, 2=Somewhat Satisfied, 3=Somewhat Dissatisfied, 4=Completely Dissatisfied
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 56 | 57
participants
  Completely Satisfied | 22 | 21
  Somewhat Satisfied | 27 | 22
  Somewhat Dissatisfied | 5 | 8
  Completely Dissatisfied | 2 | 6

49. Primary Outcome: Overall Handling Satisfaction
Description: Participant rating of satisfaction regarding handling. Collected at 4 weeks wear for both study lens pairs. 4-point Likert Scale; 1=Completely Satisfied, 2=Somewhat Satisfied, 3=Somewhat Dissatisfied, 4=Completely Dissatisfied
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 56 | 57
participants
  Completely Satisfied | 42 | 44
  Somewhat Satisfied | 12 | 11
  Somewhat Dissatisfied | 1 | 2
  Completely Dissatisfied | 1 | 0

50. Primary Outcome: Overall Vision Satisfaction
Description: Participant rating of overall satisfaction for vision. Collected at 4 weeks wear for both study lens pairs. 4-point Likert Scale; 1=Completely Satisfied, 2=Somewhat Satisfied, 3=Somewhat Dissatisfied, 4=Completely Dissatisfied
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 56 | 57
participants
  Completely Satisfied | 45 | 38
  Somewhat Satisfied | 8 | 12
  Somewhat Dissatisfied | 2 | 3
  Completely Dissatisfied | 1 | 4

51. Secondary Outcome: Binocular Visual Acuity logMAR
Description: as for outcome 3
Time Frame: 4 Weeks
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 56 | 57
logMAR | -0.052 (0.0063) | -0.047 (0.058)

52. Secondary Outcome: Surface Wetting
Description: Assessment of surface wetting by slit lamp. Collected at 4 weeks wear for both study lens pairs. 0=Non-wettable surface, 1= > 1 non-wetting area of some magnitude., 2=One non-wetting area of some magnitude, 3=Hazy surface that resolves with a blink. Typical soft lens appearance with long drying time., 4=Smooth uniformly reflective surface. Appearance of a healthy cornea (Grade 0-4 in ½ steps)
Time Frame: 4 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 56 | 57
units on a scale | 7.09 (1.84) | 6.95 (1.53)

53. Secondary Outcome: Surface Deposition
Description: Assessment of surface deposition by slit lamp. Collected at 4 weeks wear for both study lens pairs. (Grade 0-4 in 1/2 steps; 0=clean, 4=deposited)
Time Frame: 4 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 56 | 57
units on a scale | 0.58 (1.18) | 1.04 (1.65)

54. Secondary Outcome: Centration
Description: Assessment of lens centration. Collected at 4 weeks wear for both study lens pairs.. Biomicroscopy, by degree and direction in the primary position. (Optimal Centration or Not Optimal)
Time Frame: 4 Weeks
Measure: Number; unit: lenses
Units Other Than Participants: lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 55 | 57
Number analyzed (lenses) | 110 | 114
lenses
  Optimal Centration | 100 | 106
  Not Optimal Centration | 10 | 8

55. Secondary Outcome: Corneal Coverage
Description: Assessment of lens corneal coverage. Collected at 4 weeks. (Biomicroscopy; assessed in primary gaze, Normal Coverage or Not Covering)
Time Frame: 4 Weeks
Measure: Number; unit: lenses
Units Other Than Participants: lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 55 | 57
Number analyzed (lenses) | 110 | 114
lenses
  Normal Coverage | 110 | 114
  Not Covering | 0 | 0

56. Secondary Outcome: Post Blink Movement
Description: Assessment of post blink movement. Collected at 4 weeks. Assessed immediately after the blink. (Graded 0-4, 0=Insufficient, unacceptable movement, 1=Minimal, but acceptable movement, 2=Optimal movement, 3=Moderate, but acceptable movement, 4=Excessive, unacceptable movement)
Time Frame: 4 Weeks
Measure: Number; unit: units on a scale
Units Other Than Participants: lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 55 | 57
Number analyzed (lenses) | 110 | 114
units on a scale
  Movement Grade 0 | 0 | 0
  Movement Grade 1 | 8 | 11
  Movement Grade 2 | 96 | 92
  Movement Grade 3 | 6 | 9
  Movement Grade 4 | 0 | 2

57. Secondary Outcome: Push Up Test
Description: Assessment of lens tightness. Collected at 4 weeks. Digital push up test. (Continuous Scale 0-100%, 0%=Falls from cornea without lid support, 50%= Optimum, 100%= No movement)
Time Frame: 4 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 55 | 57
Number analyzed (lenses) | 110 | 114
units on a scale | 51.73 (10.80) | 52.24 (10.46)

58. Secondary Outcome: Overall Fit Acceptance
Description: Assessment of overall lens fit acceptance. Collected at 4 weeks. (0-4, 0=should not be worn, 1=borderline but unacceptable, 2=minimally acceptable, early review, 3=not perfect but OK to dispense, 4=perfect)
Time Frame: 4 Weeks
Measure: Number; unit: lenses
Units Other Than Participants: lenses
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 55 | 57
Number analyzed (lenses) | 110 | 114
lenses
  Grade 0 | 0 | 0
  Grade 1 | 0 | 0
  Grade 2 | 6 | 4
  Grade 3 | 17 | 36
  Grade 4 | 87 | 72

59. Secondary Outcome: Likelihood of Switching From Habitual Lens to Study Lens
Description: Participant likelihood of switching from their habitual lens to the study lens. Collected at 4 weeks wear for both study lens pairs. 4-point Likert Scale; 1=very likely, 2=likely, 3=unlikely, 4=very unlikely
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 56 | 57
participants
  very likely | 10 | 9
  likely | 22 | 9
  unlikely | 13 | 16
  very unlikely | 11 | 23

60. Secondary Outcome: Likelihood to Continue Wearing the Study Lens
Description: Participant likelihood of continuing wear of the study lense. Collected at 4 weeks wear for both study lens pairs. 4-point Likert Scale; 1=Very Likely, 2=Likely, 3=Unlikely, 4=Very Unlikely
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 56 | 57
participants
  Very Likely | 13 | 6
  Likely | 23 | 13
  Unlikely | 10 | 19
  Very Unlikely | 10 | 19

61. Primary Outcome: Overall Satisfaction
Description: Participant rating of satisfaction overall. Collected at 4 weeks wear for both study lens pairs. 4-point Likert Scale; 1=Completely Satisfied, 2=Somewhat Satisfied, 3=Somewhat Dissatisfied, 4=Completely Dissatisfied
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 56 | 57
participants
  Completely Satisfied | 28 | 23
  Somewhat Satisfied | 22 | 23
  Somewhat Dissatisfied | 5 | 9
  Completely Dissatisfied | 1 | 2

62. Secondary Outcome: Participant Recommendation of a Study Lens
Description: Participant most likely recommendation of which study lens to friends, family or colleagues. Collected at study exit. (Forced Choice; Study Pair 1, Study Pair 2).
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 53 | 53
participants | 31 | 22

63. Secondary Outcome: Participant Likelihood of Recommendation of a Study Lens
Description: Participant likelihood of recommending a study lens to friends. Collected at study exit. (1-4; 1=Very Unlikely, 2=Unlikely, 3=Likely, 4=Very Likely).
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 53 | 53
participants
  Very Unlikely | 6 | 12
  Unlikely | 6 | 11
  Likely | 19 | 16
  Very Likely | 22 | 14

64. Primary Outcome: Lens Preference
Description: Participant lens preference in regard for comfort, dryness, handling, vision and overall. Collected at 4 weeks. (Forced Choice; Study Pair 1, Study Pair 2).
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Comfilcon A | Lotrafilcon B
Number analyzed (Participants) | 53 | 53
participants
  Comfort | 32 | 21
  Dryness | 32 | 21
  Handling | 30 | 23
  Vision | 33 | 20
  Overall | 32 | 21

65. Primary Outcome: Lens Preference Comfort, Dryness, Vision and Overall.
Description: Participant lens preference regarding comfort, dryness, vision and overall. Collected at study exit. (Forced Choice; Study Pair 1, Study Pair 2, Habitual).
Time Frame: 4 weeks
Measure: Number; unit: participants
Groups:
- Habitual Lens: Subjects attended baseline visit wearing habitual lenses prior to dispense of study lens.
Arm/Group | Comfilcon A | Lotrafilcon B | Habitual Lens
Number analyzed (Participants) | 53 | 53 | 53
participants
  Comfort | 24 | 10 | 19
  Dryness | 23 | 11 | 19
  Vision | 23 | 10 | 20
  Overall | 22 | 10 | 21

66. Primary Outcome: Lens Preference for Handling
Description: Participant lens preference regarding handling. Collected at study exit. (Forced Choice; Study Pair 1, Study Pair 2, Habitual).
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Comfilcon A | Lotrafilcon B | Habitual Lens
Number analyzed (Participants) | 54 | 54 | 54
participants | 21 | 14 | 19

ADVERSE EVENTS:
Arm/Group | Comfilcon A | Lotrafilcon B
Serious Adverse Events (participants affected / at risk) | 1/63 | 0/63
Other Adverse Events (participants affected / at risk) | 0/63 | 0/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Comfilcon A (N=63) | Lotrafilcon B (N=63)
Peripheral Corneal Ulcer (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigators will not be permitted to publish or present at scientific meetings results obtained from the clinical study without prior written consent from the sponsor.